CLINICAL TRIAL: NCT06224530
Title: Investigating the Effect of a Single-dose of Levetiracetam on Brain Function, Chemistry and Cognitive Performance in Psychosis Risk
Acronym: LEVHIPPRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 331790; 223486/Z/21/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Psychosis
Keywords: Clinical high risk; Levetiracetam; Psychosis risk; Neuroimaging; Hippocampus; GABA; Glutamate; SV2A; Experimental medicine; Magnetic Resonance Spectroscopy; Magnetic Resonance Imaging
MeSH Terms: conditions — Psychotic Disorders | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Basic science study involving procedures with human participants. Randomised, double-blind, placebo-paired, levetiracetam versus placebo challenge before scanning. Comparison of CHR individuals (n=36) under placebo condition to baseline HC (n=33) without administration of medication.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and investigators will be blinded to the randomised order of administration of levetiracetam and placebo.
  Once screening procedures have confirmed the subject's eligibility to enter the study, a random list (i.e., of A B B A A A B B) will be created using an automated online random generator. A researcher that is not involved in the study will be responsible for randomisation and documentation. This information will then be given to the South London and Maudsley NHS Foundation Trust Pharmacy where the levetiracetam / placebo capsules will be dispensed from in visually identical capsules for blinding to the A's or B's. Only the SLaM Pharmacy contact will know what capsules were allocated to A's or B's and will keep the enrolment log blinded from the enrolment log kept by the study researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam, then Placebo (Experimental): Participants will receive two levetiracetam 250mg capsules on the first scanning visit. On the second scanning visit they will receive two 37.5mg capsules of ascorbic acid.
  Interventions: Drug: Levetiracetam; Drug: Placebo
- Placebo, then Levetiracetam (Experimental): Participants will receive two 37.5mg capsules of ascorbic acid on the first scanning visit. On the second scanning visit they will receive two levetiracetam 250mg capsules.
  Interventions: Drug: Levetiracetam; Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Single dose of 500mg levetiracetam The capsules of levetiracetam and placebo will be visibly the same.
  Other Names: Keppra
Drug: Placebo — Single dose of 75mg ascorbic acid. The capsules of levetiracetam and placebo will be visibly the same.

SUMMARY:
Background

Psychosis is a mental health condition that affects around 3 in 100 people in their lifetime. Most treatments for psychosis target a brain chemical called dopamine but they don't work for everyone and don't address many of the symptoms.

People with psychosis and people at risk of developing psychosis show differences in a part of the brain called the hippocampus, such as smaller size and increased activity. This hyperactivity may be associated with cognitive difficulties (thinking and memory).

The basis of this hippocampal hyperactivity is thought to be a deficit in excitation and inhibition of brain cells. Excitation causes brain cells to send signals more frequently, and inhibition causes cells to send signals less frequently. A balance between these signals is important for the brain, including the hippocampus, to function properly.

Approach

Levetiracetam is a medication that is widely used to treat epilepsy and which helps balance excitation-inhibition in the brain. We will use brain imaging, using Magnetic Resonance Imaging (MRI), to test if levetiracetam can help reduce hippocampal hyperactivity, alter connectivity and change levels of brain chemicals in people who are at risk of developing psychosis.

Participants (18-40 years), identified as at risk of psychosis through the Outreach and Support in South London (OASIS) teams, will attend an initial visit at the Institute of Psychiatry, Psychology & Neuroscience. This will involve questions about experiences and feelings, assessment of thinking and memory, and a blood test. They will then attend two scanning visits at the Centre for Neuroimaging Sciences, during which they will take capsules of either levetiracetam or placebo (in a randomised order) before having a 60 mins MRI scan. The MRI scan will look at blood flow to the hippocampus, resting activity, activity during a cognitive task and levels of brain chemicals.

A case-control sample of 33 healthy individuals aged 18-40 will be recruited from Greater London. We will recruit a healthy control (HC) sample to establish the presence of hippocampal dysfunction in our CHR-P group by comparing the MRI data for CHR-P under the placebo condition with that of the HC sample. The HC individuals will attend the screening visit and one scanning visit. They will not receive any medication.

Funded by the Wellcome Trust and conducted by King's College London researchers, the study spans 2-3 months per participant.

Impact

Our study will provide important evidence about how levetiracetam affects brain function, and how this relates to cognition. This knowledge may lead to innovative approaches for understanding and treating psychosis early.

DETAILED DESCRIPTION:
Can the acute administration of levetiracetam modulate hippocampal rCBF, resting-state fMRI connectivity, cognitive performance and cortical glutamatergic levels in CHR individuals?

Study Design:

Investigators will address the above research question using a randomised, double-blind, placebo-paired, within-subject crossover design on 36 participants at CHR for psychosis. The study will enrich the CHR sample and reduce heterogeneity by selecting patients who present with positive symptoms (score 3-5 on Clinical Assessment of At Risk Mental State (CAARMS) unusual thought content or non-bizarre ideas subscales), as known proxy measures of hippocampal dysfunction (Allen et al., 2018a; Modinos et al., 2018; Tregellas et al., 2014).

Previous rCBF studies including our own (Allen et al., 2016, 2018a; Percie du Sert et al., 2023) have robustly demonstrated hippocampal hyperactivity in CHR individuals compared to healthy controls. Nevertheless, the presence of hippocampal dysfunction in our CHR group will be established by comparing the MRI data for CHR under placebo condition with that of 33 healthy controls recruited from the Greater London area.

Sample:

36 individuals at CHR of psychosis 33 healthy control participants

Methodology:

CHR-P participants will undergo:

* Screening visit
* Scanning Visit 1 (under placebo/levetiracetam)
* Scanning Visit 2 (under levetiracetam/placebo)

HC participants will undergo:

* Screening visit (without blood test)
* Scanning Visit 1 (without administration of any medication)

SCREENING VISIT:

The screening visit will last approximately 2 hours (CHR-P) or 1.5 hours (HCs) and will be conducted at the IoPPN by a qualified study researcher. Procedures during this visit, except blood sampling for CHR-P and cognitive assessments, may also be conducted remotely over the telephone or video call (e.g. Microsoft Teams) in the case that a face-to-face meeting is not possible or feasible without putting participant and researcher at risk. All participants that undergo screening are logged into a screening log associated with the study by the study researcher, to which only authorized members of the research team can access (Dr Modinos and trained research workers).

- Procedures involved in the screening visit:

* Consent / capacity assessment
* Sociodemographic information, including medical, family, substance use history (including current pregnancy and breast feeding)
* Brief assessment of inclusion/exclusion criteria - including MRI safety questionnaire
* Blood sampling (CHR-P only)_
* Clinical assessment (see below)
* Cognitive assessment (see below)

Clinical assessment:

* Psychopathology will be assessed using the CAARMS.
* Anxiety and mood will be assessed using the Hamilton Anxiety and Depression Rating Scale (HAM-A/D).
* Social functioning, disability, adjustment, and interactions, and emotional empathy will be assessed using the Social and Occupational Functioning Scale (SOFAS, Global Functioning Social and Role, GF-S/R)

Cognitive assessment:

* Wechsler Adult Intelligence Scale (WAIS-III) short version (Current IQ)
* National Adult Reading Test (NART) (Premorbid IQ)
* Pattern separation task
* Cambridge Neuropsychological Test Automated Battery (CANTAB)- specific battery used for previous multi-site study PSYSCAN

Study drug / placebo (CHR only):

The study drug (500mg levetiracetam) and placebo (75mg ascorbic acid) capsules will be encapsulated, stored and dispensed by the South London and Maudsley (SLaM) NHS Foundation Trust Pharmacy. Levetiracetam / placebo capsules will be dispensed in visually identical capsules for blinding purposes.

SCANNING VISITS CHR-P

MRI scans will take place at the Centre for Neuroimaging Sciences, IoPPN. Scanning visit 1 and 2 will be identical, the only difference being the administration of either placebo or levetiracetam.

Schedule:

* 90 min Arrive at the centre
* 80 min ID, neuroimaging consent and pre-scan checklist. Basic physical examination (weight, height, blood pressure, and standard systems exam). Urine drug screen (UDS) and urine pregnancy test (for female participants).
* 60min Dose of levetiracetam or placebo administered.
* 25 min Administration of emotion recognition and spatial span tasks. T = 0 MRI scan

  * 60min End scan. Subject escorted to recovery room. Subject provided with snack and refreshment.
  * 70 min Post-scan monitoring.

Scanning Visits HCs MRI scans will take place at the Centre for Neuroimaging Sciences, IoPPN..

* 45 mins Arrive at the centre

  -- 40 mins ID, neuroimaging consent and recap of pre-scan checklist. Measurement of weight and height. UDS.
* 30 mins Administration of emotion recognition and spatial span tasks. T = 0 MRI scan

  * 60min End scan. Subject provided with optional snack and refreshment.

Emotion Recognition Task The CANTAB Emotion Recognition Task66 will be administered after the levetiracetam/placebo dose (CHR-P only) and before MRI imaging. This computer-generated paradigm measures the six basic facial emotional expressions: anger, disgust, fear, happiness, sadness and surprise. Participants are presented with computer-morphed faces expressing one emotion, with each face shown for 200 ms. Participants are then required to select the displayed emotion from the six basic emotions or choose a neutral option. The task lasts approximately 12 minutes. Outcome measures include percentage and number of correct or incorrect responses and overall response latencies, which can be analysed either across individual emotions or across all emotions.

Spatial Span Task The CANTAB Spatial Span66 assesses visuospatial working memory capacity and will be administered after the levetiracetam/placebo dose (CHR-P) and before MRI imaging. In this computerised task, participants are shown white squares on a screen, some of which briefly change colour in a variable sequence. Participants are required to select the boxes that changed colour in the same order displayed by the computer, either as shown or in reverse. The sequence ranges from two to nine boxes changing colour, with varied colour throughout. Outcome measures include span length errors, number of attempts, and latency.

MRI imaging:

Neuroimaging data will be acquired using an MRI scanner at the Centre for Neuroimaging Sciences, IoPPN. Each scanning session will involve 1 hour waiting time prior to scanning to allow for the drug to exert its effects, followed by 60 minutes of scanning:

* Scene processing task.
* Glutamate and GABA Magnetic Resonance Spectroscopy (MRS)
* Resting-State fMRI
* Arterial Spin Labelling (ASL)
* Structural MRI

Drug / Placebo Administration (CHR only):

An oral dose of levetiracetam (500 mg) or placebo (75mg ascorbic acid) will be given 1 h before the beginning of the neuroimaging acquisition. This time interval is chosen because levetiracetam has peak plasma concentration (Cmax) 1 - 1.5 hours after administration. It is rapidly and almost completely absorbed following oral administration with >95% bioavailability.

Half of the sample will be given placebo in the first experimental session and levetiracetam in the second experimental session, and the other half will be given levetiracetam in the first experimental session.

Timing of Assessments:

Scanning visit 1 must be completed within three months of the screening visit. The timing of scanning visit 2 is relative to scanning visit 1. This will result in a comparable study completion period between participants. Scanning visit 2 occurs 3 weeks +/- 1 week after scanning visit 1, to allow for complete washout. Levetiracetam has a half life of 6-8 hours in healthy adults.

Duration of study:

The study will take 24 - 36 months. Each participant will be enrolled in the study for approximately 3 months from recruitment to completion of the study (screening visit + scanning visit 1 + scanning visit 2), although note that participants will only be required to attend for a few hours for each visit.

Sample size and power calculation:

Investigators will aim to recruit 36 CHR participants to allow for potential drop out rate of 20%, aiming for at least 29 subjects with both scans complete.

There are no existing studies of rCBF or other fMRI changes with levetiracetam in CHR individuals. Studies with levetiracetam administration in participants Mild Cognitive Impairment (MCI) (n= 17) have shown that levetiracetam significantly reduced mean task-based hippocampal BOLD-fMRI activation (t = 2.537, p = 0.022) to a level that no longer significantly differed from controls (n=22)(Bakker et al., 2012).

A recent study completed by the Modinos group (unpublished data) has shown that acute diazepam administration in 24 CHR individuals significantly reduced rCBF in the right (t=-4.30, FDR-corrected p<0.001) and left hippocampus (t=-2.69, FDR-corrected p=0.015).

Multiple studies have demonstrated significantly higher hippocampal rCBF for CHR individuals compared to healthy controls (Allen et al., 2016, 2018b). Allen et al (2018) showed an effect size of 0.62 for increased rCBF in the hippocampal region of interest (ROI) in CHR compared to controls (Allen et al., 2016, 2018a). Based on this, a sample size of 29 subjects will have at least 0.90 power (alpha= 0.05, two-tailed paired t-test) to detect a significant change in rCBF.

Based on the effect size of 0.62 from Allen et al (2018), with 33 CHR participants and 33 HC we will have at least 0.80 power (alpha= 0.05, independent samples t-test) to detect a significant difference in rCBF.

These estimates are conservative as this study benefits from a within-subject crossover design, which will reduce variability and confounding, and enrichment of the sample to reduce inter-subject variability.

Image Analysis and Statistics

Hypothesis 1. CHR-P MRI scans in the placebo condition will significantly differ from MRI scans obtained from HCs.

Differences in MRI outcomes will be analysed via one-way ANOVAs, controlling for confounding variables (age, sex) as covariates of no interest in the design.

Hypothesis 2. Levetiracetam (vs placebo) will decrease hippocampal rCBF in people at CHR-P of psychosis.

rCBF data will be pre-processed using the Automatic Software for ASL Processing (ASAP) 2.0 toolbox52.

Differences in hippocampal rCBF between levetiracetam and placebo conditions will be tested using a hippocampal ROI approach, via a paired t-test (p<0.05 family-wise error corrected).

Hypothesis 3. Levetiracetam (vs placebo) will improve hippocampal resting-state functional connectivity.

Resting-state fMRI data will be analysed using a seed-based approach for the hippocampus in the CONN-fMRI Functional Connectivity toolbox53. Differences between levetiracetam and placebo will be tested using paired t-tests. Dynamic connectivity will be analysed using edge-centric analysis in Matlab54. The frequency and amplitude of co-fluctuation peaks for levetiracetam vs placebo will be compared using paired t-tests (p<0.05 family-wise error corrected).

The Amplitude of Low-Frequency Fluctuation (ALFF) analysis will be performed using the current recommended methodology. The ALFF data for levetiracetam vs placebo will be compared using paired t-tests (p<0.05 family-wise error corrected).

Hypothesis 4. Levetiracetam (vs placebo) will improve hippocampal fMRI activation during a scene processing task.

The scene processing fMRI task first level analysis will include separate regressors for scene, face and scramble conditions. For second-level analysis we will use a contrast estimating the difference in average response to scene and face, versus the scrambled condition. We will perform whole-brain analysis, and ROI analysis for the hippocampus, for levetiracetam vs placebo conditions using paired t-tests (p<0.05 family-wise error corrected). Performance on the 1-back task will be measured using mean hit rate, correct rejection rate, and reaction time for each condition. To examine differences in performance we will conduct within-subject ANOVAs on hit rate, correct rejection rate, and reaction time, with group as a within-subject factors.

Hypothesis 5. Levetiracetam (vs placebo) will decrease levels of cortical glutamatergic metabolites and increase levels of GABA.

1H-MRS data will be analysed according to current recommendations. Changes in Glx levels (glutamate + glutamine) and GABA between levetiracetam and placebo conditions will be assessed using a paired t-test (p<0.05, two-tailed).

Hypothesis 6. Levetiracetam (vs placebo) will improve accuracy and latency in an emotion recognition task.

Drug effects on emotion recognition task accuracy and reaction time will be analysed using repeated-measures ANOVA, with drug (levetiracetam, placebo) and emotion (anger, disgust, fear, happiness, sadness, and surprise) as within-subject factors. Post-hoc paired t-tests with Bonferroni corrections will be used for pairwise comparisons between the drug and placebo conditions. Significance will be set at p<0.05.

Hypothesis 7. Levetiracetam (vs placebo) will improve visuospatial working memory capacity in a spatial span working memory.

Drug effects on span length, errors, number of attempts, and latency will be analysed using repeated-measures ANOVA with drug condition as a within-subject factor. Post-hoc paired t-tests with Bonferroni corrections will be used for pairwise comparisons between the drug and placebo conditions. Significance will be set at p<0.05.

Hypothesis 8. The above neuroimaging measures are associated with changes in emotion recognition and visuospatial working memory capacity.

Multiple regression analyses will be used to examine the correlations between the changes in the neuroimaging measures (levetiracetam vs placebo) and changes in visuospatial working memory and emotion recognition performance. Significance will be set at p<0.05.

Hypothesis 9. The above neuroimaging measures are associated with baseline cognitive function, clinical symptoms and blood markers.

Pearson's correlation (Bonferroni corrected p<0.05, two-tailed) will be used to test for associations between changes in the MRI measures for levetiracetam and placebo and baseline symptom severity (CAARMS symptom scores and CANTAB cognitive performance), to determine whether those CHR-P individuals with higher symptom severity / cognitive dysfunction show a greater change in MRI measures after levetiracetam.

Pearson's correlation (Bonferroni corrected p<0.05, two-tailed) will be used to test for associations between peripheral blood markers and hippocampal rCBF, and cognitive performance.

ELIGIBILITY:
CHR-P inclusion criteria

1. Age range 18-40 years
2. Capacity to consent to participation in the study
3. Inclusion into attenuated psychosis group as assessed by the CAARMS
4. Scores 3-5 on CAARMS unusual thought content or non-bizarre ideas subscales

CHR-P exclusion criteria:

1. Past episode of psychosis
2. Current exposure to drugs with strong GABAergic or glutamatergic effects (benzodiazepines, anticonvulsants, mood stabilisers, zopiclone, zolpidem, ketamine, opiates, atomoxetine, memantine)
3. Current/recent exposure to any antipsychotic medication
4. Diagnosis of any neurological disorder, including epilepsy
5. Current pregnancy/breastfeeding
6. Severe renal impairment
7. Known allergy to levetiracetam
8. Contraindication to MRI scanning
9. IQ<70 as determined with WAIS-III
10. CHR-P individuals are not deemed to have a full-blown mental health disorder. However, in the event that a CHR-P individual is acutely ill and lacking capacity to consent, they will not be approached to take part in this study.

HC inclusion criteria

1. Age range 18-40 years
2. Capacity to consent to participation in the study

HC exclusion criteria:

1. Personal history of mental health conditions
2. Any first-degree relative with a psychotic disorder
3. Diagnosis of any neurological disorder, including epilepsy
4. Currently pregnant, breastfeeding, or trying to conceive
5. Current exposure to drugs with strong GABAergic or glutamatergic effects (benzodiazepines, anticonvulsants, mood stabilisers, zopiclone, zolpidem, ketamine, opiates, atomoxetine, memantine)
6. Current/recent exposure to any antipsychotic medication
7. Contraindication to MRI scanning
8. IQ<70 as determined with WAIS-III

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance Imaging (MRI) measure of rCBF using arterial spin labelling (ASL) in the hippocampus. | 1 hour after single dose levetiracetam vs placebo
  3D pseudo-Continuous Arterial Spin Labelling (3D-pCASL) sequence will be used to measure rCBF.

SECONDARY OUTCOMES:
Brain functional resting-state fMRI measures (including Amplitude of Low-Frequency Fluctuation (ALFF)) | 1 hour after single dose levetiracetam vs placebo
  A state-of-the-art resting-state fMRI sequence will be used to measure intrinsic activity and connectivity of the hippocampus.
Brain functional MRI activation during a scene processing task. | 1 hour after single dose levetiracetam vs placebo
  Scene processing tasks have been used before in fMRI studies with the general population and patients with early psychosis. Research has demonstrated that perceptual scene processing involves the hippocampus, and this is not just dependent on memory encoding. This task demonstrated reduced fMRI activation and increase cerebral blood volume in the anterior hippocampus of patients with early psychosis compared to controls. This task will last approximately 5 minutes.
Levels of GABAergic and glutamatergic metabolites in the anterior cingulate cortex (ACC) as measured by proton magnetic resonance spectroscopy (1H-MRS). | 1 hour after single dose levetiracetam vs placebo
  1H-MRS spectra will be acquired in the ACC using a well-established local protocol for glutamate and GABA quantification (MEGA-PRESS)
Emotion recognition performance | 30 mins after single dose of levetiracetam vs placebo and at screening visit
  The CANTAB Emotion Recognition Task will be administered after the levetiracetam/placebo dose (CHR-P only) and before MRI imaging.
Spatial Span working memory performance | 30 mins after administration of levetiracetam/placebo and at screening visit for CHR participants
  Visuospatial working memory performance as measured by the CANTAB Spatial Span working memory task measured 30mins after administration of levetiracetam/placebo, before the MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Modinos, BSc MSc PhD, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology and Neuroscience, King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No